CLINICAL TRIAL: NCT05231460
Title: Do Experience of Pain and 30-Day Surgery Outcomes Differ in Robotic Bariatric Surgery Patients Treated With Narcotic vs. Non-narcotic Pain Management Protocols?
Brief Title: Pain Management Study
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Christine Lovato, Clinical Assistant Professor, Surgery, University of Arizona
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2108122253
Record Dates: First submitted 2021-12-21; First posted 2022-02-09 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Pain, Postoperative
Keywords: Transversus Abdominis Plane (TAP) Block; Bariatric Surgery; Pain, post-operative; Analgesics, Non-Narcotic; Analgesics, Narcotic; Sleeve gastrectomy; Gastric Sleeve; Postoperative Complications
MeSH Terms: conditions — Pain, Postoperative; Bites and Stings; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Each subject will be randomized at 1:1 ratio to receive either the Narcotic Pain Regimen or the Non-narcotic Pain Regimen and will also be randomized at 1:1 ratio to receive either TAP block or no TAP block. Eligible subjects will therefore be randomized to one of four arms with approximately equal sizes:1) narcotic regimen with TAP block; 2) narcotic regimen with no TAP block; 3) non-narcotic regimen with TAP block; 4) non-narcotic regimen with no TAP block.
  The primary comparison will be between narcotic and non-narcotic regimens (arms 1 and 2 combined versus arms 3 and 4 combined). Comparison of TAP block versus no TAP block (arms 1 and 3 combined versus arms 2 and 4 combined) will performed as a secondary analysis.
Masking Description: Treating surgeon will not be blinded to randomizations. Anesthesiologist providing the Tap Block will be blinded to narcotic arm and unblinded to Tap vs No Tap. Study Coordinator will be blinded to Tap vs No Tap. Statistician will be unblinded to both groups at end of study for final analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- narcotic regimen with TAP block (Active Comparator): Patient will receive Tap Block and will be administered the Narcotic Pain Regimen post-operatively
  Interventions: Drug: Active Comparator: narcotic regimen with TAP block
- narcotic regimen with no TAP block (Active Comparator): Patient will not receive TAP block and will be administered the Narcotic Pain Regimen post-operatively
  Interventions: Drug: Active Comparator: narcotic regimen with no TAP block
- non-narcotic regimen with TAP block (Active Comparator): Patient will receive Tap Block and will be administered Non-narcotic Pain Regimen post-operatively
  Interventions: Drug: non-narcotic regimen with TAP block
- non-narcotic regimen with no TAP block (Active Comparator): Patient will not receive TAP block and will be administered Non-narcotic Pain Regimen post-operatively
  Interventions: Drug: non-narcotic regimen with no TAP block

INTERVENTIONS:
Drug: Active Comparator: narcotic regimen with TAP block — Patient will receive Tap Block to 15ml of 0.5% Ropivacaine and will be administered the following Narcotic Pain Regimen post-operatively:
  * PO Oxycodone 5mg, 10mg q4h for moderate and severe pain
  * IV Dilaudid 1mg q3h for breakthrough pain
  Arms: narcotic regimen with TAP block
Drug: Active Comparator: narcotic regimen with no TAP block — Patient will not receive TAP block and will be administered the following Narcotic Pain Regimen post-operatively:
  * PO Oxycodone 5mg, 10mg q4h for moderate and severe pain
  * IV Dilaudid 1mg q3h for breakthrough pain
  Arms: narcotic regimen with no TAP block
Drug: non-narcotic regimen with TAP block — Patient will receive Tap Block to 15ml of 0.5% Ropivacaine and will be administered the following Non-narcotic Pain Regimen post-operatively:
  * Toradol 15mg q6h
  * Tylenol 1000mg q8h
  * Gabapentin 100mg three times a day
  Arms: non-narcotic regimen with TAP block
Drug: non-narcotic regimen with no TAP block — Patient will not receive TAP block and will be administered the following Non-narcotic Pain Regimen post-operatively:
  * Toradol 15mg q6h
  * Tylenol 1000mg q8h
  * Gabapentin 100mg three times a day
  Arms: non-narcotic regimen with no TAP block

SUMMARY:
This study aims to better understand the role that narcotic vs. non-narcotic multimodal pain management play in patients' pain following bariatric surgery (Laproscopic Surgery and Robotic Assisted Surgery). Participation in this study will last approximately 90 days following surgery. During that 90 day period, participants will be asked to report pain and nausea every 4 hours to a study coordinator or nurse while they are recovering in the hospital. Following discharge from the hospital patients will be asked to report pain, nausea, and any medical changes 7 days, 30 days, and 90 days from surgical date.

The procedures and medications used in this study are FDA approved medical therapies and are part of Standard of Care for this population. This study aims to therapeutically investigate efficacy of the proposed pain management regimens. The procedures and individual medications are not the subject of research as they are considered routine well established and documented interventions for obesity and the treatment of post operative pain.

DETAILED DESCRIPTION:
The majority of patients who undergo surgery will require treatment for the management of acute post-surgical pain. The use of narcotics after elective surgical procedures has contributed to the current opioid epidemic. Striking the right balance of treatment and use of narcotics vs. non-narcotic medications is at a crucial juncture in surgery.

Post-surgical pain influences a patient's perception of quality of care, physical recovery, and length of stay. The threat of poor postoperative pain control is a fear of many patients who will have a surgical procedure. The post- operative pain regimen is traditionally chosen by the operating surgeon rather than in a shared decision-making model where patients are educated about choice and participate in management. This is one of many factors influencing use of medications for post-operative pain. If a patient develops longer term, chronic postsurgical pain it may lead to disability and diminish quality of life, increase healthcare utilization, increase healthcare costs, and result in loss of productivity.

Morbid obesity is a global epidemic that increases the risk of developing related complications such as cardiac failure, type 2 diabetes, hypertension, hyperlipidemia, degenerative joint disease with the development of chronic pain and decreased mobility, and sleep apnea. In 2013 and 2014, 50% of the population had or had been affected by obesity, defined as a BMI ≥30mg/kg2. An established and effective treatment for weight loss is elective bariatric surgery.

Laparoscopic bariatric surgery (>90% of cases) is associated with less postoperative pain than open surgery, however, opioids are still used frequently for analgesia. Opioid analgesia comes with many side effects including nausea, constipation, risk of postoperative ileus, hypopnea, hypoxemia, delayed ambulation and mortality. This patient population is at increased risk for hypoventilation and narcotic related post-operative complications.

In the BUMCP department of bariatric surgery, we began employing a post-operative multimodal pain control protocol in November of 2017 and noticed improvement in pain control, declining levels of nausea and a decrease in the length of stay with our patient population. All medications and surgical interventions are considered approved standard of care in surgery. Previous studies have shown that employing a multimodal pain control protocol, even intraoperatively, influences postoperative pain control, nausea, emesis as well as chronic postoperative pain. In mid-2018 we began offering patients tap blocks which we believe have offered patients more consistent post- operative pain control.

Postsurgical pain control is imperative as it influences a patient's quality of care and life, recovery, and length of stay. Poor pain control can not only lead to increased healthcare utilization/costs, whereas use of opioid analgesia comes with side effects including nausea, constipation, risk of postoperative ileus, hypopnea, hypoxemia, delayed ambulation, mortality, and the increased possibility of long-term narcotic addiction. In the population that suffers from obesity it is desirable to reduce the narcotics being used as they are at increased risk for hypoventilation and post-operative complications. The BUMCP bariatric surgery department began employing a post-operative multimodal pain control protocol and noticed improvement in pain control, a decrease in perioperative morbidity from narcotic use and a decreased length of stay in the elective patient population undergoing primary bariatric surgery. This study will contribute to our knowledge of whether a non-narcotic, multi-modal post-operative pain management protocol is equivalent, if not superior in multiple facets compared to narcotic use.

Objectives

Study Hypothesis:

The use of a multi-modal, non-narcotic pain management regimen in postoperative bariatric patients will have equivalent, if not superior, postoperative outcomes compared with patient receiving narcotic pain management regimen. Those patients receiving a TAP block will have better pain control in the first 24 hours post-op.

Primary outcome measure:

Patient reported postoperative pain using the Wong Baker Faces pain scale (mean of all reported scores till the earlier of discharge and 24 hours postoperative).

Secondary outcomes measures:

* Postoperative nausea numerical rating scale (0-5)
* Length of time before subject can complete 200 feet of ambulation post-op
* Hospital length of stay
* Readmissions for pain control up to 30-day postoperatively (as binary Yes/No and also as a count variable)

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic or Robotic Sleeve Gastrectomy bariatric surgery scheduled electively from the BUMCP Bariatric Clinic
* BMI>35kg/m2
* Patient of Principal Investigator or Co-Investigator
* 18 years or older

Exclusion Criteria:

* Chronic Pain Management on narcotics at New Patient visit or placed on narcotics prior to surgery
* Re-operative bariatric surgery procedures
* Admitted to the ICU after surgery
* Unable to walk 200ft
* Allergic to narcotics, steroids, or other medications used in the protocol
* Use of insulin to treat diabetes
* Chronic Kidney Disease - stage 4 or greater
* Significant hepatic disease
* Carries a diagnosis of Pulmonary Hypertension
* Carries a diagnosis of Congestive Heart Failure
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | discharge or 24 hours postoperative, whichever is first
  Patient reported postoperative pain using the Wong Baker Faces pain scale. The scale shows a series of six faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable. Based on the faces and written descriptions, the patient chooses the face that best describes their level of pain.

SECONDARY OUTCOMES:
Postoperative nausea | post-operative until patient discharge or up to 90 days, whichever comes first
  Postoperative nausea defined by numerical rating scale (0-5)
200 foot ambulation | post-operative until patient discharge or up to 90 days, whichever comes first
  Length of time before subject can complete 200 feet of ambulation post-op
Hospital length of stay | post-operative until patient discharge or up to 90 days, whichever comes first
  Patient's length of stay in the hospital
Readmissions | up to 30-day postoperatively
  Readmissions for pain control

CONTACTS AND LOCATIONS:
Locations (1):
- Banner University Medical Center Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be retained for future use. Data will not be shared with collaborating entities nor sold/shared with pharmaceutical companies